CLINICAL TRIAL: NCT00944138
Title: Randomized 8-week Pilot Study of Relaxation Methods for Weight Loss in Adults With Chronic Kidney Disease
Brief Title: 8-week Pilot Study of Relaxation for Weight Loss in Adults With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Holly Kramer, Edward Hines Jr. VA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMISE#0001
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
Keywords: Obesity; meditation; chronic kidney disease
MeSH Terms: conditions — Obesity; Renal Insufficiency, Chronic

ARMS (2):
- Mindful meditation (Experimental): Participants assigned to the mindful meditation plus standard care arm will receive individualized instruction on mindful meditation at the time they are randomized to this arm. The participants will be led through a 20 minute relaxation exercise. They will then be led through a brief eating exercise where they will be instructed to eat the food very slowly and pay attention to how the food tastes and the sensations of swallowing the food. This is done to enhance the person's awareness of what and how they are eating and enhance their intuitive sense of satiety. Finally, they will receive an MP3-player with several relaxation instructional audios loaded on the MP3 player.
  Interventions: Behavioral: Relaxation methods
- Music for relaxation (Active Comparator): Participants assigned to the control arm will receive the dietary counseling and will be told that relaxation can help reduce appetite. However, techniques to relax will not be taught. Instead, participants will be encouraged to sit quietly listening to music (of their choice) every day for 20 minutes. Participants assigned to the standard care arm will receive an MP3-player and will be given a choice of selection of music that they can load on their MP3 player (classical music, country music, jazz, etc.).
  Interventions: Behavioral: Relaxation methods

INTERVENTIONS:
Behavioral: Relaxation methods — Relaxation methods will include mindful meditation techniques for the intervention and listening to music for the control arm

SUMMARY:
Obesity plays a causal role for kidney disease incidence and progression. Moderate weight loss reduces the high metabolic demands on the kidney and decreases proteinuria in both diabetic and non-diabetic nephropathies. However, maintaining behavioral changes for weight loss is very challenging, and common chronic kidney disease (CKD) co-morbidities such as decreased exercise capacity only compound this difficulty. Moreover, no weight loss medications have been adequately tested in adults with CKD and most are contraindicated in this population. Mindful meditation or "mindfulness" in addition to other relaxation techniques may help adults lose weight by interrupting learned behavior, curbing compulsive eating, and reducing stress and appetite. Although mindful meditation and other relaxation techniques have gained the attention of the mainstream media for obesity treatment, scientific data on its efficacy remain limited. Due to the short duration of this study, substantial weight loss in any participant is not expected. Instead, the primary purpose of this study is to examine the feasibility of a randomized controlled trial of mindful meditation relaxation techniques combined with standard care compared to standard care alone for the treatment of obesity among Veterans with CKD.

ELIGIBILITY:
Inclusion Criteria:

* receive medical care at the Hines VA CKD clinics.
* Presence of chronic kidney disease defined as an estimated glomerular filtration rate < 60 ml/min/1.73 m2 BSA or a spot urine albumin/creatinine ratio ≥ 30 mg/g
* BMI ≥ 35 kg/m2 or a waist circumference ≥ 102 (40 inches) and ≥ 88 cm (35 inches) in men and women, respectively.

Exclusion Criteria:

* Inability to give informed consent
* inability to come to VA for two group sessions
* inability to listen to an MP3 player using headphones

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
weight, waist circumference, measures of stress and mood and overall satisfaction | 8 nweeks

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States